CLINICAL TRIAL: NCT04288713
Title: Soliris to Stop Immune Mediated Death In Covid 19 Infected Patients. A Trial of Distal Complement Inhibition.
Brief Title: Eculizumab (Soliris) in Covid-19 Infected Patients
Acronym: SOLID-C19
Status: Available | Type: Expanded Access
Sponsor: Hudson Medical (Other)
Responsible Party: Principal Investigator, Thomas Pitts, M.D., Thomas C Pitts, M.D., Hudson Medical
Other Study IDs: COVID19
Record Dates: First submitted 2020-02-27; First posted 2020-02-28 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Coronavirus
Keywords: Covid19; Soliris; Eculizumab; Covid-19; Complement; Immunomodulation; ARDS; Adult respiratory distress syndrome; Coronavirus; Corona Virus
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Respiratory Distress Syndrome | interventions — eculizumab

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Drug: Eculizumab — A distal complement inhibitor.

SUMMARY:
Covid-19 has spread rapidly throughout the world causing widespread panic, death, and injury. While this virus is the provocateur, it is often the patient's own disproportionate immune response which deals the most devastating (and often fatal) damage. A specific part of the immune system, known as the complement, has been shown to cause such damage in other types of coronaviruses. In the SOLID-C19 study, Soliris (Eculizumab) will be used to modulate the activity of the distal complement preventing the formation of the membrane attack complex. By modulating this portion of the immune response, mortality can be halted while the patient has time to recover from the virus with supportive medical care.

DETAILED DESCRIPTION:
Recorded Endpoints:

* Mortality
* Time in the ICU
* Time on a ventilator

Administrative:

An Emergency FDA IND must be submitted (FDA form 3926) for each patient.

Subsequent to approval the primary investigator will obtain an authorization letter from Alexion Pharmaceuticals.

Implementation:

Prior to dosing the patient must receive ceftriaxone IV and this must be continued during the entire duration of therapy (vaccination will be mentioned shortly and is the only exception to prophylactic antibiotic coverage). If there is a clinical reason why the patient cannot receive Ceftriaxone (allergy, supply, etc) then an alternative prophylactic antibiotic covering Neisseria meningitis must be given for the duration of therapy. The SeroB and Quadrivalent meningococcal vaccines can be given if the duration of antibiotic therapy becomes unsafe or unfeasible. In that case, antibiotic therapy should be withdrawn no sooner than 2 weeks after vaccination with both meningococcal vaccines (see ACIP guidelines in complement deficient patients). It is preferred that vaccination is avoided while the patient is acutely ill and that prophylactic antibiotics are used as meningococcal vaccination can upregulate the immune system possibly worsening the patient's condition.

Standard dosing protocol - Eculizumab 900mg IV every 7 days. Eculizumab is given IV over 30 minutes without the need of a pump (although one can be used if available).

Supplemental doses of eculizumab can be given if clinically warranted at the discretion of the investigator and clinical team.

The team should perform Murray scores daily for the first 72 hours THEN every other day unless a change is deemed necessary by the attending physician. (table 2)

Complement blood levels should be drawn every 72 hours. They may be drawn sooner if there is clinical inquiry which would affect clinical decision making and/or after a dose of Eculizumab is given.

The duration of therapy is at the discretion of the clinical team and investigator.

Follow up at day 7, 14, and 28 after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Confirmed Covid-19 infection
* ARDS
* ICU patient

Exclusion Criteria:

* Active Neisseria infection.
* Concomitant enrollment in another experimental/off-label immunosuppressive therapy trial.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

REFERENCES:
- [Background] Gralinski LE, Sheahan TP, Morrison TE, Menachery VD, Jensen K, Leist SR, Whitmore A, Heise MT, Baric RS. Complement Activation Contributes to Severe Acute Respiratory Syndrome Coronavirus Pathogenesis. mBio. 2018 Oct 9;9(5):e01753-18. doi: 10.1128/mBio.01753-18. PMID 30301856